CLINICAL TRIAL: NCT04859179
Title: Prenatal Carrier Screening for Spinal Muscular Atrophy Among Thai Pregnant Women
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Chayada Tangshewinsirikul, Division of Maternal-Fetal Medicine, Department of Obstetrics and Gynecology, Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Mahidol University
Other Study IDs: COA. MURA2020/1420
Record Dates: First submitted 2021-03-26; First posted 2021-04-26 (Actual); Last update posted 2021-04-26 (Actual); Status verified 2021-04

CONDITIONS: Spinal Muscular Atrophy
Keywords: spinal muscular atrophy; prenatal screening
MeSH Terms: conditions — Muscular Atrophy, Spinal

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Months
Biospecimen Retention: Samples With DNA — blood, plasma and DNA
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Spinal muscular atrophy (SMA) prenatal carrier screening is recommended by American College of Medical Genetics (ACMG) and American College of Obstetrics and Gynecology (ACOG). However, in Thailand, there are no standard protocol for SMA prenatal carrier screening.

DETAILED DESCRIPTION:
Spinal muscular atrophy (SMA) is one of the most common neuromuscular autosomal recessive disorders. The incidence is about 1:10,000 livebirths. There are 5 subgroups base on onset of symptoms and clinical severity. Type 1 is the most severe type which age of onset is 6 months old and life expectancy is less than 1-2 years. SMA carrier frequency is approximately 1/40-1/60. Molecular genetic testing to detect copies number of SMN1 gene is possible with as high as 95% detection rate. Since 2008, American College of Medical Genetics (ACMG) and American College of Obstetrics and Gynecology (ACOG) recommended SMA preconceptional and prenatal carrier screening in general population. In Thailand, there are no standard protocol for SMA prenatal carrier screening.

ELIGIBILITY:
Inclusion Criteria:

* Maternal age > 18 years
* Singleton pregnancy
* Gestational age ≤ 14 weeks

Exclusion Criteria:

* Refuse to participate the research trial

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: All pregnant women who came to antenatal care clinic at Ramathibodi Hospital, Mahidol University
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-03-10 (Actual); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Rate of acceptance of prenatal carrier screening for spinal muscular atrophy | 12 months
  Rate of acceptance of prenatal carrier screening for spinal muscular atrophy among pregnant women seeking prenatal care

SECONDARY OUTCOMES:
Factors associated rate of acceptance of prenatal carrier screening for spinal muscular atrophy | 12 months
  Factors associated rate of acceptance of prenatal carrier screening for spinal muscular among pregnant women seeking prenatal care
Copies number of SMN1 and SMN2 genes in pregnant women | 12 months
  Copies number of SMN1 and SMN2 genes in pregnant women among individuals who accepted carrier screening
Carrier frequency among individuals who accepted carrier screening | 12 months
  Screen positive rate or rate of having 1 copy of SMN1 among individuals who accepted carrier screening
Pregnant women's attitudes toward spinal muscular atrophy and carrier screening | 12 months
  After genetic counseling, pregnant women's attitudes toward spinal muscular atrophy and carrier screening will be evaluated by validated questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Chayada Tangshewinsirikul, Principal Investigator — Ramathibodi Hospital, Mahidol University
Locations (1):
- Faculty of Medicine, Ramathibodi Hospital, Mahidol University, Ratchathewi, Bangkok, Thailand